CLINICAL TRIAL: NCT00004079
Title: A Phase I Trial of Sarcosinamide Nitrosourea (SarCNU) in Patients With Solid Tumors
Brief Title: Sarcosinamide Nitrosourea in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00028; 99-046; U01CA062490 (NIH); CDR0000067290 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-12-10; First posted 2003-04-09 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 2-((((2-chloroethyl)nitrosoamino)carbonyl)amino)propanamide

ARMS (1):
- Treatment (SarCNU) (Experimental): Patients receive oral sarcosinamide nitrosourea (SarCNU) on days 1, 5, and 9. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of SarCNU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: SarCNU; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: SarCNU — Given PO
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of sarcosinamide nitrosourea in treating patients who have metastatic or unresectable solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of an oral formulation of SarCNU given on an every 4th day times three schedule (days 1, 5, 9).

II. Establish an appropriate oral dose of SarCNU for phase II clinical trials. III. Identify the dose-limiting toxicities (DLTs) of SarCNU. IV. Determine the oral bioavailability of SarCNU. V. Characterize the plasma pharmacokinetics of SarCNU.

SECONDARY OBJECTIVES:

I. Determine whether SarCNU undergoes metabolic N-demethylation to generate reactive isocyanate species that have been implicated in BCNU pulmonary toxicity.

II. Evaluate response to treatment with SarCNU in patients with measurable or evaluable disease.

III. Attempt to establish pharmacodynamic relationships for response and/or toxicity.

OUTLINE: This is a dose-escalation study.

Patients receive oral sarcosinamide nitrosourea (SarCNU) on days 1, 5, and 9. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SarCNU until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 4-5 weeks posttreatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented malignancy, which is either metastatic or inoperable, for which there is no known curative or standard palliative therapy, or all standard therapeutic approaches have failed
* Patients with leukemia or primary CNS malignancies are excluded; patients with metastatic disease to the CNS, who are not receiving anticonvulsants, including phenytoin, carbamazepine, phenobarbital, primidone, and felbamate, and who have reasonable expectation of surviving long enough to receive two cycles of therapy, are eligible
* Life expectancy of 2 months or longer
* ECOG performance status of 0-2
* Pretreatment laboratory data, obtained within 14 days of study entry, must meet the following criteria:
* ANC >= 1,500 /mm^3
* Platelets >= 100,000 /mm^3
* SGOT =< 2.5-times upper limit of normal
* SGPT =< 2.5-times upper limit of normal
* Total bilirubin =< upper limit of normal
* Creatinine =< 1.5 mg/dl
* Creatinine CL >= 60 ml/min (measured 24hr) if creatinine > 1.5 mg/dl
* DLCO >= 80% predicted
* At least 4 weeks since last receiving radiotherapy or chemotherapy and complete recovery from previous treatment related toxicity
* No prior treatment with a nitrosourea or with bleomycin
* No enzyme inducing anticonvulsant agents
* At least 2 weeks since major surgery
* Patients must not have uncontrolled serious medical or psychiatric illness
* Women of childbearing potential must not be lactating or pregnant, because of the proven teratogenicity of other agents of this class; a negative pregnancy test has to be obtained within 2 weeks of entry; both fertile males and females must use adequate contraception upon entry into the study
* Patients must have given signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1999-08; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
MTD | 28 days
Pharmacokinetics: plasma concentration-time profiles of SarCNU | Days 1 and 9 of course 1: 5, 15, 20, 30, and 45 min; 1, 2, 3, 4, and 6 hr
  Analyzed by nonlinear least squares regression using WinNonlin (Scientific Consulting, Inc.). Final values of the iterated parameters in the best-fit equations describing the plasma profiles will be used to calculate all pharmacokinetic terms according to standard equations. Mean values of the pharmacokinetic parameters will be calculated at each dose and subject to appropriate statistical tests for the existence of dose-dependent trends.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Eder, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States